CLINICAL TRIAL: NCT06813677
Title: Innsbruck Health Promotion Program
Acronym: INNHEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VASCage GmbH (Other)
Collaborators: Oroboros Instruments (Unknown); Med-El Corporation (Industry); Tirol Kiniken GmbH (Other); Österreichische Gesundheitskasse (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: C_2_A.2-0062_012
Record Dates: First submitted 2025-01-13; First posted 2025-02-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Assessment of Vascular Health Risk Factors
Keywords: Life's Essential 8; PBMC; Cardiovascular health; Quality of Life; Mitochondrial function; Hearing impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health promotion arm (Experimental): Over a time period of 12 months participants will receive regular newsletters as part of the health promotion program, informing them about vascular health promotion opportunities in the region. At the end of the study participants are provided with tailored guidance on further optimizing their vascular health to reduce individual risks of stroke and heart attack.
  Interventions: Other: In-person health promotion

INTERVENTIONS:
Other: In-person health promotion — The results from the initial pre-baseline examination are reviewed during the baseline visit to identify potential risk factors related to the Life's Essential 8 (LE8). Based on these findings, participants receive personalized recommendations to enhance their vascular health and information on local vascular health promotion resources. Additionally, participants receive bi-monthly motivational newsletters designed to support ongoing vascular health improvements.

SUMMARY:
The primary goal of this single-centre. single-arm, unblinded, pre-post interventional study is to evaluate whether a one-time health assessment and intervention affects the overall vascular health evaluated through the Life's Essential 8 overall vascular health score.

Secondary goals of this study are, among others:

* to describe incidence and prevalence of vascular risk-factors and behaviours
* to explore prevalence and associations of health and disease in the general population with special focus on cardiovascular risk, cardiovascular diseases, markers of vascular health, signs and (prodromal) symptoms of neurodegeneration as well as psychosocial factors
* to explore the prevalence of hearing disorders in the general population
* to collect voice and speech samples to identify novel biomarkers that correlate to vascular health and/or hearing status

DETAILED DESCRIPTION:
Cardio- and cerebrovascular diseases are the leading cause of death and disability globally, underscoring the need for primary prevention, especially given that 80% of stroke patients in Tyrol had untreated risk conditions prior to their stroke.

The American Heart Association (AHA) and the American Stroke Association (ASA) identify eight factors that have a fundamental influence on vascular health, collectively known as "Life's Essential 8" or "LE8." The LE8 includes blood pressure, blood sugar, LDL cholesterol, BMI (Body Mass Index), as well as physical activity, sleep, a balanced diet, and avoiding nicotine products.

The INN.HEALTH study aims to evaluate the impact of a single health examination with counseling, supplemented by bi-monthly motivational newsletters, on improving vascular health over one year among a large cohort of Tyrolean adults. For this purpose, 1000 participants (500 men, 500 women) from various age groups are recruited and comprehensively characterized in terms of their demographic information and clinical profiles.

During the initial baseline pre-examination (study visit 1), blood, urine and stool samples are collected, and selected participants receive an actigraphy device for monitoring activity patterns. Additionally, participants complete self-administered questionnaires about their lifestyle habits. Two weeks post pre-examination (baseline, study visit 2) physical assessments and cognitive and sensory tests are performed. Based on these results the participant's health status in relation to the LE8 factors is assessed and the reduction of identified risk factors is discussed in a counseling session. If certain findings require further clarification, participants are referred to a specialist for further evaluation and treatment.One year after the initial examinations, participants are scheduled for two additional appointments: the first one (study visit 3) is identical to the initial baseline pre-examination, the second one marks the final examination (study visit 4), and is identical to baseline.

Over the 12 months between study visits 2 and 3 participants receive regular newsletters as part of the health promotion program, informing them about vascular health promotion opportunities in the region.

In the final consultation at the end of the final examination visit, participants receive a comprehensive assessment of which aspects of their lifestyle have significantly changed over the past year. Participants are then provided with tailored guidance on further optimizing their vascular health to reduce individual risks of stroke and heart attack.

Secondary objectives of this study include analyzing changes in quality of life, medication compliance, healthcare usage, vascular and cognitive health, as well as identifying risk factors and early markers for neurodegenerative disease, with data collected and periodically reviewed long-term. The study also seeks to establish a regional cohort with a biobank for future research on vascular health, aging, and mitochondrial function, and to explore the feasibility of incorporating hearing screenings into routine health exams

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent of subject
* Main area of residence in Innsbruck and Innsbruck-Land

Exclusion Criteria:

* People who are suspended upon a court order or upon other legal processes or are accommodated according ot the Hospitalization Act, or for whom a custodian is appointed (or appointment is inititated)
* Persons with impaired power of judgement
* Persons who are currently engaged in military or community service

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Life's Essential 8 overall cardiovascular health | Pre-baseline examination (day 0)
  Changes in Life's Essential 8 (LE8) overall cardiovascular health metric between baseline and follow-up examination.
  Scores are categorized as low (0-49), moderate (50-79), or high (80-100). A higher LE8 score indicates better cardiovascular health and is associated with a lower risk of cardiovascular diseases (CVD) and mortality.

SECONDARY OUTCOMES:
Changes in individual components of Life's Essential 8 - Diet | At pre-baseline examination (day 0) and at follow-up pre-examination (12 +/- 2 months after baseline)
  Assessment of change in diet using the Food Frequency Questionnaire
Changes in individual components of Life's Essential 8 - Diet | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in diet using the Mediterranean Eating Pattern for Americans (MEPA) Score. Score minimum 0, score maximum 100. A higher score indicates a diet closely aligned with the mediterranean eating pattern.
Changes in individual components of Life's Essential 8 - Physical activity | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in physical activity with focus on amount and intensity of physical activity
Changes in individual components of Life's Essential 8 - Nicotine Exposure | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in smoking status
Changes in individual components of Life's Essential 8 - Body weight | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in body weight (body mass index, kg)
Changes in individual components of Life's Essential 8 - Blood lipids | At pre-baseline examination (day 0) and at follow-up pre-examination (12 +/- 2 months after baseline)
  Assessment of change in blood lipid levels: triglyceride (mmol/L), cholesterol (all, mmol/L)
Changes in individual components of Life's Essential 8 - Body glucose | At pre-baseline examination (day 0) and at follow-up pre-examination (12 +/- 2 months after baseline)
  Assessment of change in blood glucose levels: fasting glucose (mg/dL, mmol/L)
Changes in individual components of Life's Essential 8 - Blood glucose | At pre-baseline examination (day 0) and at follow-up pre-examination (12 +/- 2 months after baseline)
  Assessment of changes in blood glucose levels: HbA1c (%)
Changes in individual components of Life's Essential 8 - Blood pressure | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in blood pressure (systolic/diastolic, mmHg)
Changes in individual components of Life's Essential 8 - Sleep | At pre-baseline examination (day 0) and at follow-up pre-examination (12 +/- 2 months after baseline)
  Assessment of change in sleep quality using the Pittsburgh Sleep Quality Index
Changes in individual components of Life's Essential 8 - Sleep | At baseline (day 14) and at follow-up (2 weeks after follow-up pre-examination)
  Assessment of change in sleep habits

CONTACTS AND LOCATIONS:
Overall Officials: Dr.med. Lukas Mayer-Süß, PhD, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University Innsbruck - Department of Neurology, Innsbruck, Austria